CLINICAL TRIAL: NCT01037465
Title: ROS Signaling in Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Naomi M Hamburg, Principal Investigator, Boston University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-26547
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Disease
Keywords: endothelium; cell signaling; N-acetylcysteine; reactive oxygen species
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Active Comparator): N-acetylcysteine
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine
  Arms: N-acetylcysteine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The vascular endothelium (inner lining of cells in blood vessels) normally prevents vasospasm and thrombosis by producing nitric oxide and other regulatory substances. In patients with atherosclerosis, endothelial function is impaired. Excess production of reactive oxygen species (free radicals) contribute to endothelial dysfunction in atherosclerosis, and some prior studies have shown a beneficial effect of antioxidant treatment on endothelial function in patients with coronary artery disease. On the other hand, reactive oxygen species may be required for normal endothelial function and antioxidant supplements failed to show a benefit in large clinical trials. The effect of antioxidant treatment on endothelial function in healthy subjects is unknown. The present study will test the hypothesis that scavenging reactive species might reduce endothelium-dependent vasodilation in healthy subjects.

The study is a randomized, double-blind, placebo-controlled crossover study. Participants will receive 2.4 grams of oral NAC or similar-appearing placebo during the first visit, and then will cross over to the alternative treatment (NAC or placebo) for the second and final visit. We will examine endothelial function before and after treatment on each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Male and Female subjects.
2. Age range: 21-65 years old.
3. Disease status: No acute, chronic, or debilitating medical condition or use of prescribed medications.
4. Willingness and ability to provide written informed consent and the ability to understand, to participate and to comply with the study requirements.

Exclusion Criteria:

1. Women with a positive urine beta HCG pregnancy test and lactating women.
2. Blood pressure greater than 140/90 mmHg; serum LDL cholesterol greater than 160 mg/dl; fasting blood sugar greater than 110 mg/dl.
3. History of any cigarette smoking within one year of the study.
4. Clinical history of any acute, chronic, or debilitating medical condition, including liver disease and peptic ulcer disease.
5. Treatment with an investigational new drug within the last 30 days.
6. History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03-26 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 4 hours

SECONDARY OUTCOMES:
Blood markers of antioxidant capacity | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hamburg, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No